CLINICAL TRIAL: NCT03858829
Title: Development and Validation of a Scale to Measure Fear of ACTivity in Patients With Coronary Artery Disease - (Fact-CAD)
Brief Title: Development and Validation of a Scale to Measure Fear of ACTivity in Patients With Coronary Artery Disease
Acronym: Fact-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25901600/893
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; physical activity; cardiac rehabilitation; validation studies; psychometrics
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fear of movement scale (Experimental)
  Interventions: Other: Psychometric analysis

INTERVENTIONS:
Other: Psychometric analysis — Psychometric analysis

SUMMARY:
Low motivation to exercise is one of the barriers to participation in cardiac rehabilitation. Fear of activity after a cardiac event is associated with low levels of physical activity. This study aimed to develop and validate a scale to measure fear of activity in patients with coronary artery disease.

DETAILED DESCRIPTION:
Low motivation to exercise is one of the barriers to participation in cardiac rehabilitation. Fear of activity after a cardiac event is associated with low levels of physical activity. This study aimed to develop and validate a scale to measure fear of activity in patients with coronary artery disease. A scale for Fear of ACTivity in patients with CAD (Fact-CAD) was created through semi-structured focus group interviews with patients. Face and content validity of Fact-CAD was verified. The scale was applied to 250 patients who had myocardial infarction, coronary artery bypass grafting or percutaneous coronary intervention within the last 12 months. Psychometric analysis included model fit, unidimensionality, reliability, local dependency, differential item functioning and external construct validity. Analyses were performed using the Rasch Analysis Model.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had myocardial infarction, coronary artery bypass grafting or percutaneous coronary intervention within the last 12 months.

Exclusion Criteria:

* Acute cardiac event within the last month
* Attendance to cardiac rehabilitation
* İnability to read and understand,
* İnability to ambulate or unwillingness to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
A scale for fear of activity | baseline
  Each item is scored by a 5-point likert scale (4= always, 3= mostly, 2= sometimes, 1= seldom, 0= never). The scale is bi-directional; seven items 1, 5, 9, 13, 17, 19 and 21 are positively designed and their scores are inversely scored (0= always, 1= mostly, 2= sometimes, 3= seldom, 4= never). Total score is calculated by summing the scores of each item. Higher scores indicate the severity of fear of activity.

SECONDARY OUTCOMES:
Nottingham Health Profile | baseline
  It contains 38 items that address pain, physical mobility, emotional reactions, energy, social isolation, and sleep dimensions. Higher scores indicate worse quality of life.
Beck Depression Inventory | baseline
  This is a 21-item self-report questionnaire evaluating the presence and severity of depressive symptoms in the vegetative, emotional, cognitive and motivational domains. Scores of each item ranges from 0 to 3, higher scores mean higher risk of depression.
Beck Anxiety Inventory | baseline
  Each item is rated on 4-point scale ranging from 0 to 3. Four items are related to anxiety mood, four items related to specific fears and fourteen items are related to physiological aspects of anxiety such as autonomic hyperactivity. Higher scores indicate higher levels of anxiety.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozyemisci-Taskiran O, Demirsoy N, Atan T, Yuksel S, Coskun O, Aytur YK, Tur BS, Karakas M, Turak O, Topal S. Development and Validation of a Scale to Measure Fear of Activity in Patients With Coronary Artery Disease (Fact-CAD). Arch Phys Med Rehabil. 2020 Mar;101(3):479-486. doi: 10.1016/j.apmr.2019.09.001. Epub 2019 Sep 25. PMID 31562874